CLINICAL TRIAL: NCT06554587
Title: Evaluation of the Performance of the Glycoscore Biomarkers for the Detection of Clinically Significant Prostate Cancer
Brief Title: Investigation of Three Biomarkers for the Detection of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Medtechtomarket Consulting Ltd (Industry)
Collaborators: GlycoscoreDx Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: M2M-GLYCOSCORE-01
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples retained from consenting patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected prostate cancer or on active surveillance: Diagnostic tests to measure three separate biomarkers in blood taken from patients pre-biopsy to assess the diagnostic performance of the biomarkers in detecting clinically significant prostate cancer (Gleason score ≥7)
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis: Enzyme-linked immunosorbent assay (ELISA)

INTERVENTIONS:
Diagnostic Test: Laboratory Biomarker Analysis: Enzyme-linked immunosorbent assay (ELISA) — Measurement of the plasma concentration of ST6GAL1, GCNT1 and GALNT7 biomarkers in patients suspected of having prostate cancer or on active surveillance

SUMMARY:
GlycoScore Dx Limited, a diagnostics company based in the United Kingdom have identified three glycoproteins, that showed promise as biomarkers of prostate cancer in initial validation studies. The purpose of this study is to further evaluate the sensitivity and specificity of the GlycoScore biomarkers for the detection of clinically significant prostate cancer. Sensitivity and specificity will be determined for each marker, combinations of the three markers and combinations of the GlycoScore biomarkers with PSA (prostate specific antigen). The results from this study will be used to identify the most suitable biomarker/biomarkers for use in developing a GlycoScore test.

This is a prospective, non-interventional study using venous blood samples taken from patients with suspected prostate cancer or on active surveillance, attending the hospital Urology department for a transperineal biopsy.

DETAILED DESCRIPTION:
Worldwide, prostate cancer is the most commonly diagnosed cancer in men and the fifth leading cause of cancer death in men. This amounted to 1,414,249 newly diagnosed cases and 375,000 deaths worldwide yearly from this disease in 2020. Globally, prostate cancer is the most commonly diagnosed cancer in more than fifty percent of countries (112 of 185). It presents a significant clinical burden in terms of volume and as a diagnostic challenge.

The initial diagnosis of prostate cancer relies on the detection of PSA (prostate specific antigen) in patient blood. While PSA is relatively good at identifying prostate cancer, PSA levels can be elevated for reasons other than cancer (giving a false positive result). Two thirds of men with a raised PSA level don't have prostate cancer meaning that many men undergo unnecessary & invasive follow up procedures, such as tissue biopsy. Prostate biopsies place a huge burden on both healthcare systems, and individuals with suspected prostate cancer. They are painful, can lead to complications, infections and in extreme circumstances, death.

Therefore, the poor specificity of the PSA test, combined with the disparate natural histories of many prostate cancers has limited its utility as a screening tool.

A combination of clinical and pathological features, such as the tumour grade (Gleason score or Gleason Grade Group), combined with clinical examination (digital rectal examination), MRI (magnetic resonance imaging) and isotope bone scan are commonly used to determine the aggressiveness and curability of tumours with radical treatment. PSA measurement is used as part of this assessment but, as other factors can influence PSA levels, it cannot be used to assess risk or guide treatment in isolation.

There remains an unmet clinical need for a better screening and diagnostic test for prostate cancer. Such a test must also be able to differentiate between early, low-risk cancers that do not require radical treatment and more aggressive tumours where radical treatment is preferable. By identifying which patients have a clinically significant risk of prostate cancer we believe our test could provide a solution to both.

The GlycoScore immunoassays detect the three biomarkers - 'glycosyltransferase enzymes' in patient blood (GALNT7, ST6GAL1 and GCNT1) which are linked to key tumour-associated glycans (types of sugars on cell walls) using an ELISA (enzyme-linked immunosorbent assay-based platform).

Initial studies conducted by Newcastle University using RUO (research use only) ELISA kits showed a significant correlation between prostate cancer and the three biomarkers ST6GAL1, GCNT1 and GALNT7. Extensive research and development work has been carried out developing custom antibody pairs and antigens for inclusion in our ELISA kit, as well as to optimize buffers and other components.

The purpose of this study is to obtain fresh patient blood samples to further evaluate the three biomarkers ST6GAL1, GCNT1 and GALNT7 for their ability to identify clinically significant prostate cancer, either alone, as a combination of the biomarkers or in combination with the PSA (measurement obtained at Medtechtomarket) using our in-house developed ELISA assays and a CE-marked PSA ELISA test kit.

Diagnostic accuracy for participants with prostate cancer will be determined by comparison with biopsy results, and for participants without prostate cancer, comparison with mpMRI (multi-parametric magnetic resonance imaging) and biopsy results.

Assessment of the correlation between the GlycoScore biomarker results with the full range of biopsy Gleason scores/Gleason Grade group/CPG grade (Cambridge Prognostic Group) will allow an assessment of the prognostic value of the GlycoScore test and its potential use in the clinical management of prostate cancer.

Patients attending the hospital for a transperineal prostate biopsy who are either being investigated for suspected prostate cancer or are undergoing active surveillance for previously diagnosed prostate cancer will be asked to consent to take part in the study. Patients will be asked to consent to have a small sample of blood taken before the biopsy and for study investigators to have access to their final diagnosis. The blood sample will be sent to Medtechtomarket Laboratories for measurement of the biomarkers and PSA. Patients will also be asked to consent to an additional tube of blood to be taken (from the same blood draw) and the urine sample, which is routinely taken before the biopsy to be sent to the Liverpool University Biobank for future use in research studies.

137 male patients aged 18 years and above will be recruited for the study which is expected to take 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years and over
* The patient is being investigated for suspected prostate cancer or is on active surveillance
* The patient is able to give consent to take part in the study

Exclusion Criteria:

* A patient who has already taken part in the study
* A patient with an active urinary tract infection
* The patient has a prior diagnosis of any other cancer or is receiving any cancer treatment (including ADT)
* The patient is currently or within the last 4 months enrolled on another study involving an investigational medicinal product

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients referred to the secondary care (urology clinic) for transperineal biopsy for the investigation of suspected prostate cancer or patients undergoing active surveillance
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
An evaluation of the diagnostic performance of the GlycoScore biomarkers for the detection of clinically significant prostate cancer (Gleason score of ≥7). | Pre-biopsy (one time point)
  A comparison of calculated sensitivity, specificity and positive and negative predictive values for clinically significant prostate cancer for the following:
  Each biomarker, alone and in combination with PSA (measured on from the same blood sample using a CE-marked assay)
  Each possible combination of GlycoScore biomarkers, alone and in combination with PSA
  The reference method for diagnosis of prostate cancer will be biopsy, and the reference method for identifying patients who do not have cancer will be by a combination of mpMRI and/or biopsy.

SECONDARY OUTCOMES:
Establishment of a 'GlycoScore' algorithm | Pre-biopsy (one time point)
  Establish an algorithm for calculating a 'GlycoScore' that converts the assay results from the optimal combination of biomarkers into a score that indicates the likelihood that a patient has clinically significant prostate cancer (Gleason score of ≥7).
An evaluation of the ability of the calculated 'GlycoScore' to distinguish between individual Gleason scores and grade groups | Pre-biopsy (one time point)
  Correlation between the calculated 'GlycoScore' from each sample and Gleason score and grade groups at biopsy
An evaluation of the ability of the calculated 'GlycoScore' to distinguish between CPG groups 1 to 5 (Cambridge Prognostic Group classification) | Pre-biopsy (one time point)
  Correlation between the calculated 'GlycoScore' from each sample and the Cambridge Prognostic Group classification
A comparison of the diagnostic performance of the GlycoScore biomarkers (with and without PSA) against the performance of the hospital PSA test alone for the detection of clinically significant prostate cancer (Gleason score of ≥7). | Pre-biopsy (one time point)
  A comparison of calculated sensitivity, specificity and positive and negative predictive values for clinically significant prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Lazarowicz, FRCS(Urol), Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roddam AW, Duffy MJ, Hamdy FC, Ward AM, Patnick J, Price CP, Rimmer J, Sturgeon C, White P, Allen NE; NHS Prostate Cancer Risk Management Programme. Use of prostate-specific antigen (PSA) isoforms for the detection of prostate cancer in men with a PSA level of 2-10 ng/ml: systematic review and meta-analysis. Eur Urol. 2005 Sep;48(3):386-99; discussion 398-9. doi: 10.1016/j.eururo.2005.04.015. PMID 15982797
- [Background] Catalona WJ, Hudson MA, Scardino PT, Richie JP, Ahmann FR, Flanigan RC, DeKernion JB, Ratliff TL, Kavoussi LR, Dalkin BL, Waters WB, MacFarlane MT, Southwick PC. Selection of optimal prostate specific antigen cutoffs for early detection of prostate cancer: receiver operating characteristic curves. J Urol. 1994 Dec;152(6 Pt 1):2037-42. doi: 10.1016/s0022-5347(17)32300-5. PMID 7525995
- [Background] Johnston E, Pye H, Bonet-Carne E, Panagiotaki E, Patel D, Galazi M, Heavey S, Carmona L, Freeman A, Trevisan G, Allen C, Kirkham A, Burling K, Stevens N, Hawkes D, Emberton M, Moore C, Ahmed HU, Atkinson D, Rodriguez-Justo M, Ng T, Alexander D, Whitaker H, Punwani S. INNOVATE: A prospective cohort study combining serum and urinary biomarkers with novel diffusion-weighted magnetic resonance imaging for the prediction and characterization of prostate cancer. BMC Cancer. 2016 Oct 21;16(1):816. doi: 10.1186/s12885-016-2856-2. PMID 27769214
- [Background] Tuck MK, Chan DW, Chia D, Godwin AK, Grizzle WE, Krueger KE, Rom W, Sanda M, Sorbara L, Stass S, Wang W, Brenner DE. Standard operating procedures for serum and plasma collection: early detection research network consensus statement standard operating procedure integration working group. J Proteome Res. 2009 Jan;8(1):113-7. doi: 10.1021/pr800545q. PMID 19072545
- [Background] Flahault A, Cadilhac M, Thomas G. Sample size calculation should be performed for design accuracy in diagnostic test studies. J Clin Epidemiol. 2005 Aug;58(8):859-62. doi: 10.1016/j.jclinepi.2004.12.009. PMID 16018921
- See also: Prostate cancer: diagnosis and management - current UK NICE guidelines — https://www.nice.org.uk/guidance/ng131
- See also: Current NICE guidelines - Evidence review covering the definition of clinically significant prostate cancer, page 17 — https://www.nice.org.uk/guidance/ng131/evidence/d-diagnosing-and-identifying-clinically-significant-prostate-cancer-pdf-6779081777

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT06554587/Prot_SAP_003.pdf